CLINICAL TRIAL: NCT02724189
Title: The Evaluation of MyPreOp© (Online Pre-assessment Tool) Over a Conventional Nurse Led Pre-assessment Clinic: a Pilot and Feasibility Study.
Brief Title: The Evaluation of MyPreOp, an Online Preoperative Assessment Tool
Status: Terminated | Type: Observational
Why Stopped: Lack of logistic capabilities at the study site
Sponsor: Michelle Cole (Other)
Responsible Party: Sponsor-Investigator, Michelle Cole, Perioperative Medicine Fellow, University College London Hospitals
Organization: University College London Hospitals (Other)
Other Study IDs: 15/0795
Record Dates: First submitted 2016-03-21; First posted 2016-03-31 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Focus of Study: The Safety of an Online Pre-assessment Tool
Keywords: electronic pre-assessment; preoperative assessment

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients attending the preoperative assessment clinic: Patients in preoperative assessment clinic
  Interventions: Device: MyPreOp assessment; Other: Nurse led assessment

INTERVENTIONS:
Device: MyPreOp assessment — MyPreOp is an online preoperative assessment programme created by a medical software company called Ultramed.
Other: Nurse led assessment — Standard practise is where patients undergo a face to face preoperative assessment led by a qualified nurse specialising in this field.
  Other Names: Standard

SUMMARY:
This pilot study will intend to assess the feasibility and acceptability of MyPreOp (online pre-operative assessment tool). The study will aim to assess the quality of the MyPreOp assessment in comparison to standard practice of a nurse led face to face assessment. The investigators will also assess the acceptability of MyPreOp amongst patient participants and staff participants.

DETAILED DESCRIPTION:
MyPreOp is a patient online pre-assessment tool that has been developed as a means of an alternative to the current existing model of a nurse led pre-assessment service.

This pilot study will intend to assess the feasibility and acceptability of MyPreOp. The study will primarily evaluate the quality of the MyPreOp assessment in comparison to standard practice of a nurse led assessment. The investigators will also assess the acceptability of MyPreOp amongst patient participants and pre-assessment nurses and anaesthetists.

Participants will be recruited directly from the pre-assessment clinic. Consenting participants will alternate undergoing either the MyPreOp assessment or the nurse assessment first. Participants will complete the MyPreOp assessment on a computer device at the hospital. Participants will also complete a nurse led pre-assessment process as per standard practice. Following the completion of both the MyPreOp assessment and the nurse assessment, participants will be asked to complete a satisfaction questionnaire about their experience of using MyPreOp, together with further questions about their home internet access, usage and their preference of electronic or nurse led assessments.

Similarly pre-assessment nurses will review a random sample of MyPreOp assessments and complete a questionnaire about their views of the MyPreOp assessment summary and recommended actions.

The MyPreOp assessments will be compared with the nurse assessments through an independent adjudication process. Nominated adjudicators will be Consultant Anaesthetists with regular clinical duties in the pre-assessment clinic. Adjudicators will not be blinded with respects to the assessments so that the manner in which the patient data is presented can also be compared as well as the data itself. Adjudicators will assess the performance of the MyPreOp assessment in two domains, medical history and recommended investigations, and assign them into graded categories of over or under assessment, with or without clinical significance.

ELIGIBILITY:
Inclusion Criteria:

* All patients due to see a pre-assessment nurse on that day
* Read and able to write English
* Lucid patients with mental capacity

Exclusion Criteria:

* Patients unable to understand spoken or written English.
* Not able to see a pre-assessment nurse on the same day
* Patients too unwell or confused to be able to complete the questionnaire.
* Patient refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study group will be taken from a single centre. The patient population will be patients being assessed prior to general, gynaecological, urological and orthopaedic surgery. The investigators selected this population as they represent a diverse sample of patients of both genders with a varying range of ages and co-morbidities for both ambulatory and inpatient surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The event rate of MyPreOp assessments that are judged as under assessments that would affect perioperative management following an adjudication review | Through study completion,an average of 6 months

SECONDARY OUTCOMES:
Percentage of participants requiring assistance to complete MyPreOp | Through study completion,an average of 6 months
The median time taken for a nurse assessment of the MyPreOp summaries | Through study completion,an average of 6 months
  This will be collected from the nurse questionnaire data ie the nurse would report the time taken to assess the MyPreOp summaries. The investigators will not be directly measuring the time.
Patient satisfaction | Through study completion,an average of 6 months
  Qualitative analysis of patient satisfaction when using MyPreOp. The data will be extracted from the patient satisfaction questionnaire.
Nurse satisfaction | Through study completion,an average of 6 months
  Qualitative analysis of nurse satisfaction when evaluating the MyPreOp summaries. The data will be extracted from the nurse satisfaction questionnaire.
Anaesthetist satisfaction | Through study completion,an average of 6 months
  Qualitative analysis of anaesthetic satisfaction when evaluating the MyPreOp summaries. The data will be extracted from the anaesthetic satisfaction questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ramani Moonesinghe, FRCA MD(Res), Study Chair — Director UCL/UCLH Surgical Outcomes Resource Centre, Consultant Anaesthetics and Intensive Care Medicine, UCLH Honorary Lecturer

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to publish anonymised study results on the Surgical Outcome Research Centre website. http://www.uclsource.com/